CLINICAL TRIAL: NCT00766116
Title: A Phase I/II Trial of the Combination 5-azacitidine and Gemtuzumab Ozogamicin Therapy for Treatment of Relapsed AML
Brief Title: Combination 5-azacitidine and Gemtuzumab Ozogamicin Therapy for Treatment of Relapsed Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Celgene Corporation (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, Edward Ball, Professor of medicine, University of California, San Diego
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 090516
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1 Dose Level 1 (Experimental): 5-Azacitidine, Gemtuzumab ozogamicin
  75 mg/m^2 5-Aza 2 days then GO at 3 mg/m^2
  Interventions: Drug: 5-Azacitidine; Drug: Gemtuzumab ozogamicin
- Phase 1 Dose Level 2 (Experimental): 5-Azacitidine, Gemtuzumab ozogamicin
  75mg/m^2 5-Aza for 4 days then GO at 6 mg/m^2
  Interventions: Drug: 5-Azacitidine; Drug: Gemtuzumab ozogamicin
- Phase I Dose Level 3 (Experimental): 5-Azacitidine, Gemtuzumab ozogamicin
  75 mg/m^2 5-Aza for 6 days then GO at 6 mg/m^2
  Interventions: Drug: 5-Azacitidine; Drug: Gemtuzumab ozogamicin
- Phase 2 Dose Level 1 (Experimental): 5-Azacitidine, Gemtuzumab ozogamicin
  75 mg/m^2 5-Aza for 6 days then GO at 6 mg/m^2
  Interventions: Drug: 5-Azacitidine; Drug: Gemtuzumab ozogamicin

INTERVENTIONS:
Drug: 5-Azacitidine — Given in cohorts of 3 starting with 2 doses of 5-azacitidine. The doses of 5-azacitidine will be escalated to 4 and then 6 doses if the dose escalation rules permit.
  Other Names: Vidaz
Drug: Gemtuzumab ozogamicin — Mylotarg given 2 times over 2 weeks
  Other Names: Mylotarg

SUMMARY:
This study will test an experimental combination of the drugs Mylotarg and 5-azacitidine in the hopes of finding a treatment that may be effective against Acute Myeloid Leukemia that has come back after treatment.

DETAILED DESCRIPTION:
In the Phase I portion of the study patients with a diagnosis of AML who have relapsed disease will be treated with an assigned number of doses of 5 azacitidine followed by Mylotarg administered two times over two weeks

In the Phase II portion of the study patients will be treated with the dose of 5azacitidine determined to be safe in the Phase I portion of the study followed by Mylotarg.

A sample of blood or bone marrow will be obtained prior to initiation of treatment and another sample obtained after treatment with 5-azacitidine but before Mylotarg and the samples will be tested in the laboratory to determine response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Relapsed AML
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2, and life expectancy > 3 months
* ≥ 18 years old
* Previously untreated for current AML relapse
* Adequate organ function
* Written informed consent

Exclusion Criteria:

* Pregnant or breast-feeding women
* Growth factors that support platelet or white cell number or function must not have been administered within the past 7 days
* Currently receiving another investigational drug
* Currently receiving other anti-cancer agents
* Uncontrolled infection
* HIV positive
* Received previous therapy with either Mylotarg or 5-azacitidine

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2014-09-26 (Actual); Study Completion 2014-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward D Ball, MD, Principal Investigator — UCSD
Locations (3):
- United States (3):
  - UCSD Moores Cancer Center, La Jolla, California
  - Stanford University, Stanford, California
  - Northside Hospital/BMTGA, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: 5-Azacitidine, Gemtuzumab ozogamicin
  5-Azacitidine: A = given in cohorts of 3 starting with 2 doses of 5-azacitidine. The doses of 5-azacitidine will be escalated to 4 and then 6 doses if the dose escalation rules permit
  Gemtuzumab ozogamicin: M = Mylotarg given 2 times over 2 weeks
Period: Overall Study
Arm/Group | Treatment
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: MTD was the maximum number of 5-azacitadine doses (75mg/m2) at which fewer than 1/3 of patients experienced a DLT during cycle 1 of therapy based on CTCAE Version 3.0. In the phase I portion, we assessed 3 dose levels of azacitidine starting on day 1, with 6, 4, and 4 patients in cohort 1, 2, and 3, respectively. We identified no dose-limiting toxicities and identified the phase 2 dose as 75 mg/m2 of 5-azacitadine for 6 days.
Time Frame: up to 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Cohort 1: 5-Azacitidine, Gemtuzumab ozogamicin- Phase 1 Dose Cohort 1: 75 mg/m2 daily for 2 days
- Phase 1 Cohort 2: 5-Azacitidine, Gemtuzumab ozogamicin- Phase 1 Dose Cohort 1: 75 mg/m2 daily for 4 days
- Phase 1 Cohort 3: 5-Azacitidine, Gemtuzumab ozogamicin- Phase 1 Dose Cohort 1: 75 mg/m2 daily for 6 days
Arm/Group | Phase 1 Cohort 1 | Phase 1 Cohort 2 | Phase 1 Cohort 3
Number analyzed (Participants) | 6 | 4 | 4
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Response to the Combination Treatment of Mylotarg With 5-azacitidine
Time Frame: Hematologic and Cytogeneic Response to treatment will be assessed when evaluated at the time the ANC has reached 1000/mm3 for three consecutive days, assessed up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 36
Participants | 36

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 20/50
Other Adverse Events (participants affected / at risk) | 44/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=50)
Pneumonia (Infections and infestations) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
fever/pneumonia (Infections and infestations) | 1 (1)
Gram (-) Rods (Infections and infestations) | 1 (1)
nausea, vomiting, abdominal pain (Gastrointestinal disorders) | 1 (1)
Hospitalized with syncopal event with intraventricular hemorrhage. (Infections and infestations) | 1 (1)
Hypotension second to Mylotarg infusion (Cardiac disorders) | 1 (1)
Infection documented/ relapsed AML (Infections and infestations) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 11 (13)
Refractory platlets (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
SIRS (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=50)
Febrile Neutropenia (Blood and lymphatic system disorders) | 38 (46)
Gram Positive Infections (Infections and infestations) | 7
Gram Negative Infections (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 5 (8)
Abnormalities in liver function tests (Blood and lymphatic system disorders) | 5 (5)
Mucositis (Gastrointestinal disorders) | 6 (6)
SIRS/Sepsis (Infections and infestations) | 5 (5)
Weakness (General disorders) | 5 (15)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Electrolyte abnormalities (Blood and lymphatic system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes